CLINICAL TRIAL: NCT03586726
Title: A Single-Center, Non-Randomized, Open-Label, One-Sequence, Two-Period Within-Subject Study to Investigate the Effect of Rifampicin on the Pharmacokinetics of Multiple Doses of Balovaptin In Healthy Volunteers
Brief Title: A Study to Investigate the Effect of Rifampicin on the PK of Multiple Doses of Balovaptin In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WP40608; 2018-001783-40 (EudraCT Number)
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — balovaptan; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balovaptan + Rifampicin (Experimental): Participants received the study drugs in 2 periods. There was a minimum of a 14-day to a maximum of a 21-day washout between the last dose in Period 1 and the first dose in Period 2.
  Interventions: Drug: Balovaptan; Drug: Rifampicin

INTERVENTIONS:
Drug: Balovaptan — In Period 1, balovaptan was administered alone as a once daily (qd) dose on Days 1 to 10.
  In Period 2, balovaptan was administered as a qd dose on Days 7 to 16.
Drug: Rifampicin — In Period 2, 600 mg of rifampicin will be administered alone as a qd dose from Day 1 to Day 6, and as a qd dose on Days 7 to 16.

SUMMARY:
This study was a single-center, non-randomized, open-label, one-sequence, two-period, within-subject study to investigate the effects of multiple doses of rifampicin on the PK and safety of multiple doses of balovaptan in healthy subjects. The study was conducted at 1 site in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, urinalysis, and serology.
* Body Mass Index of 18 to 30 kg/m2, inclusive.
* For women of childbearing potential: agreement to use at least 2 acceptable contraceptive methods during the treatment period and for 90 days after the last dose of study drug.
* For men: agreement to use contraceptive measures, and agreement to refrain from donating sperm until 90 days after the last dose of study drug.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator.

Rifampicin-related Exclusion Criteria:

* Subjects diagnosed, or suspected of having porphyria, and subjects with first-degree relatives diagnosed, or suspected of having porphyria.
* Known hypersensitivity to rifampicin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pra International Group B.V, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derks MGM, Wandel C, Young A, Bolt SK, Meyenberg C. Open-Label Assessment of the Effects of Itraconazole and Rifampicin on Balovaptan Pharmacokinetics in Healthy Volunteers. Adv Ther. 2020 Nov;37(11):4720-4729. doi: 10.1007/s12325-020-01491-y. Epub 2020 Sep 15. PMID 32935287

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balovaptan + Rifampicin
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Balovaptan
Description: Cmax is the observed peak analyte concentration obtained directly from the experimental data without interpolation, expressed in concentration units.
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: The Pharmacokinetic (PK) analysis population consisted of all subjects who received at least one dose of balovaptan. Participants were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
ng/mL
  Balovaptan (Period 1) | 94.2 (33.4)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 12.9 (22.8)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for M2 Metabolite
Description: as for outcome 1
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
ng/mL
  Balovaptan (Period 1) | 22.0 (22.7)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 8.09 (20.5)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for M3 Metabolite
Description: as for outcome 1
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
ng/mL
  Balovaptan (Period 1) | 49.6 (26.4)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 10.9 (23.2)

4. Primary Outcome: Area Under the Plasma Concentration Curve From Time 0 to 24 Hours (AUC0-24) for Balovaptan
Description: AUC0-24 is the area under the plasma concentration-time curve from time 0 to 24 hours post dose.
Time Frame: Day 10 and 11 of Period 1; Day 16 and 17 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
ng.h/mL
  Balovaptan (Period 1) | 1000 (29.6)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 67.0 (16.3)

5. Primary Outcome: Area Under the Plasma Concentration Curve From Time 0 to 24 Hours for M2 Metabolite
Description: AUC0-24 is the area under the plasma concentration-time curve from time 0 to 24 hours post dose.
Time Frame: Day 10 and 11 of Period 1; Day 16 and 17 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
ng.h/mL
  Balovaptan (Period 1) | 448 (22.7)
  Balovaptan + rifampicin (Period 2) | 149 (21.9)

6. Primary Outcome: Area Under the Plasma Concentration Curve From Time 0 to 24 Hours for M3 Metabolite
Description: AUC0-24 is the area under the plasma concentration-time curve from time 0 to 24 hours post dose.
Time Frame: Day 10 and 11 of Period 1; Day 16 and 17 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
ng.h/mL
  Balovaptan (Period 1) | 844 (20.8)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 110 (13.3)

7. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to 21 days postdose
Population: The safety analysis population consisted of subjects who received at least one dose of balovaptan.
Measure: Number; unit: Percentage
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Percentage | 94

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for Balovaptan
Description: Tmax is the first observed time to reach peak analyte concentration obtained directly from the experimental data without interpolation, expressed in time units.
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Hour
  Balovaptan (Period 1) | 1.00 [0.50 to 1.10]
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 1.00 [0.50 to 1.02]

9. Secondary Outcome: Time to Maximum Observed Plasma Concentration for M2 Metabolite
Description: as for outcome 8
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Hours
  Balovaptan (Period 1) | 2.50 [0.00 to 16.00]
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 3.00 [1.50 to 12.00]

10. Secondary Outcome: Time to Maximum Observed Plasma Concentration for M3 Metabolite
Description: as for outcome 8
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour(s)
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Hour(s)
  Balovaptan (Period 1) | 1.00 [0.50 to 4.00]
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 1.00 [1.00 to 4.00]

11. Secondary Outcome: Metabolite to Parent Ratio for M2 Metabolite Based on AUC0-24
Time Frame: Day 10 and 11 of Period 1; Day 16 and 17 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Ratio
  Balovaptan (Period 1) | 0.430 (32.3)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 2.14 (14.8)

12. Secondary Outcome: Metabolite to Parent Ratio for M2 Metabolite Based on Cmax
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Ratio
  Balovaptan (Period 1) | 0.225 (30.9)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 0.606 (20.7)

13. Secondary Outcome: Metabolite to Parent Ratio for M3 Metabolite Based on AUC0-24
Time Frame: Day 10 and 11 of Period 1; Day 16 and 17 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Ratio
  Balovaptan (Period 1) | 0.872 (16.6)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 1.70 (6.9)

14. Secondary Outcome: Metabolite to Parent Ratio for M3 Metabolite Based on Cmax
Time Frame: Day 10 of Period 1 and Day 16 of Period 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Balovaptan + Rifampicin
Number analyzed (Participants) | 16
Ratio
  Balovaptan (Period 1) | 0.545 (16.5)
  Balovaptan + rifampicin (Period 2): number analyzed (Participants) | 15
  Balovaptan + rifampicin (Period 2) | 0.873 (9.0)

ADVERSE EVENTS:
Time Frame: Up to 21 days postdose (15 November 2018).
Groups:
- BALOVAPTAN+RIFAMPICIN: In Period 1, balovaptan was administered alone as a once daily (qd) dose on Days 1 to 10.
  In Period 2, balovaptan was administered as a qd dose on Days 7 to 16.
  In Period 2, 600 mg of rifampicin was administered alone as a qd dose on Days 7 to 16.
Arm/Group | BALOVAPTAN+RIFAMPICIN
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BALOVAPTAN+RIFAMPICIN (N=16)
Headache (Nervous system disorders) | 6 (11)
Dizziness (Nervous system disorders) | 4 (5)
Head discomfort (Nervous system disorders) | 1 (3)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2)
Chromaturia (Renal and urinary disorders) | 12 (14)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (3)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (7)
Nightmare (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stifness (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Catheter site pain (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-06-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT03586726/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03586726/SAP_001.pdf